CLINICAL TRIAL: NCT04554303
Title: A 12 Weeks, Multi-center, Randomized, Open Label, Active Control, Phase IV Clinical Trial to Compare Evaluated Improvement of Edema Index, Safety and Efficacy of Amlodipine Versus S Amlodipine in Patients With Essential Hypertension
Brief Title: Comparing Safety and Efficacy of Amlodipine Verses S Amlodipine in Patients With Essential Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Collaborators: Korea University Guro Hospital (Other); Dt&Sanomedics (Industry)
Responsible Party: Sponsor
Other Study IDs: AG-C1908
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-09

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Amlodipine; S-Amlodipine; Hypertension; Blood Pressure; Edema
MeSH Terms: conditions — Essential Hypertension; Hypertension; Edema | interventions — levamlodipine; Amlodipine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- S-amlodipine treatment group: Patients with essential hypertension, who satisfies all criteria listed in eligibility section are randomly assigned, after a wash-out period of at least two weeks.
  Interventions: Drug: S-amlodipine 2.5mg
- Amlodipine treatment group: Patients with essential hypertension, who satisfies all criteria listed in eligibility section are randomly assigned, after a wash-out period of at least two weeks.
  Interventions: Drug: Amlodipine 5mg

INTERVENTIONS:
Drug: S-amlodipine 2.5mg — Oral administration, 1 tablet per day
  Other Names: Levotension Tab.
  Groups: S-amlodipine treatment group
Drug: Amlodipine 5mg — Oral administration, 1 tablet per day
  Other Names: Norvasc Tab.
  Groups: Amlodipine treatment group

SUMMARY:
As a third-generation dihydropyridine calcium channel blocker (CCB), Amlodipine is mainly used in a single therapy or combined therapy for hypertension or angina.

Edema, one of the most common side effects of dihydropyridine CCB formulations, may lead to drug control or discontinuation of drugs.

This clinical study intends to assess the safety and efficacy of S-amlodipine, which is assessed to be superior to Amlodipine in the aspects of antihypertensive effect and side effects, in edema of patients with essential hypertension.

DETAILED DESCRIPTION:
1. Clinical Study Design

   - In this clinical study, Part 1 is conducted as a preliminary study on 10 subjects at a single center, and based on the results of Part 1, the sponsor and the principal investigator determine whether to proceed with Part 2. With Part 2 as the multicenter main study conducted on the remaining 70 subjects, 80 subjects in total have been planned for Part 1 and Part 2.
2. Interim analysis

   - The interim analysis is conducted when the study on 10 subjects at a Part 1 single center has been completed; the analysis is made on all endpoints planned for this clinical study.
3. Clinical study methods - During screening, subjects who have voluntarily signed the Informed Consent Form are tested for eligibility to this clinical study.

After a wash-out period of at least two weeks, subjects who satisfy the inclusion/exclusion criteria are randomly assigned to two groups (S-amlodipine group, Amlodipine group). Thereafter, the subjects are enrolled and orally administered with the investigational product once a day for 12 weeks, during which they receive a total of five visits for tests conducted for assessment of efficacy and safety.

(In case of confirmed eligibility without administration of contraindications, the wash-out period may be omitted and Visits 1 and 2 may be paid on the same day)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension and diagnosed with stage 1-2 hypertension in accordance with the 2019 Korean Society of Hypertension criteria (SBP ≥ 140 mmHg or DBP ≥ 90 mmHg)
2. Where a subject and his/her spouse (partner) have agreed to use medically acceptable contraceptives in the following during participation in this clinical study:

   * Use of intrauterine device with proven failure rate of pregnancy;
   * Simultaneous use of blocking contraception and spermicide;
   * Has had a vasectomy;
   * Has had a salpingectomy, tubal ligation, or hysterectomy;
3. Those who have made voluntary decisions to participate in this clinical study and have consented to the Informed Consent Form in writing;
4. Those who are able to understand and follow instructions and participate throughout the entire clinical study

Exclusion Criteria:

1. Patients with uncontrolled, high-risk hypertension (SBP≥180mm Hg and DBP≥110mm Hg);
2. Those who have a history of secondary hypertension and any history of suspected secondary hypertension (aortic congestion, hyperaldosteronism, renal artery stenosis, Cushing's disease, chromaffinoma, polycystic renal disease, etc.);
3. Those who fall under one or more of the following items that may cause edema without underlying diseases:

   * Those who have been diagnosed with myocardial infarction or heart failure within 6 months of screening;
   * Those who have been diagnosed with a cerebrovascular accident (CVA) within 6 months of screening;
   * Patients with renal failure requiring dialysis or those with edema caused by renal dysfunction (renal salt retention);
   * Those who have uncontrolled diabetes (HbA1c> 10.0%) or diabetic edema;
   * Patients with severe liver dysfunction or edema caused by liver disease (cirrhosis);
   * Other patients with hypothyroidism, proteinuria, and problems at the joint or ankle joint
4. Those who have cerebrovascular disease, unstable angina, or transient ischemic attack, or those who have had coronary artery bypass graft or coronary angioplasty;
5. Patients who may develop edema by concomitant drugs at screening:

   * Drugs that constrict intrarenal blood vessels (e.g. nonsteroidal anti-inflammatory drugs, cyclosporine, etc.);
   * Drugs that dilate arterioles (e.g. vasodilators, etc.);
   * Drugs that increase sodium reabsorption in the kidneys (e.g. steroids, etc.);
   * Drugs that damage capillaries (e.g. interleukin-2, etc.);
   * Glitazone-based drugs for diabetes
6. Those who show hypersensitive reaction* to the investigational product;
7. Those who are taking the following drugs that may cause drug interactions:

   * Drugs that may change the plasma concentration of amlodipine [e.g. CYP3A4 inducers (e.g. rifampicin, St. John's wort (Hypericum perforatum), etc.);
   * Drugs that may increase the antihypertensive action [e.g. other antihypertensives (calcium channel blockers, beta blockers, ACEi, ARB, alpha blockers, diuretics, nitroglycerin), tricyclic antidepressants (amitriptyline, desipramine, imipramine, nortriptyline, protriptyline, trimipramine, etc.), nitrate formulation, baclofen, pioglitazone, sildenafil, etc.];
   * Systemic corticosteroids (fluocinolone, triamcinolone), etc.: Local application allowed;
   * Drugs that may increase the inhibitory action of muscle contraction [e.g. antiarrhythmics (amiodarone, quinidine, etc.);
   * Drugs that may cause ventricular spasms (e.g. intravenous administration of dantrolene and verapamil);
   * Drugs that may increase the risk of hypotension [e.g. CYP3A4 inhibitors (clarithromycin), etc.]
8. Patients in a state of chronic inflammation requiring chronic anti-inflammatory treatment;
9. Those who have participated in other interventional clinical studies within 6 months of screening;
10. Those who have been diagnosed as having malignant tumors within 5 years of screening;
11. Those who showed clinically significant abnormal results in electrocardiogram and laboratory tests at screening;
12. Those who are pregnant or lactating, or have been confirmed as being pregnant through the Urine HCG test;
13. Those who have been judged to be inappropriate to participate in the clinical study by the principal investigator or subinvestigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ordinary patients with essential hypertension who visits the medical institution participating in this study, and volunteers to enroll in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-05-23 (Estimated); Study Completion 2022-05-23 (Estimated)

PRIMARY OUTCOMES:
The variance in edema index [Extracellular water (ECW) / total body water (TBW)] using Inbody measurement between groups at week 12, compared to the baseline. | Edema indexs (ECW/TBW) are measured at week 4, 8, 12 of treatment.
  Descriptive statistics (number of observation subjects, mean, standard deviation, median, minimum, maximum) are summarized by treatment group. Depending on whether there is a difference in the variance between treatment groups (S-amlodipine group, Amlodipine group) that satisfies the normality assumption, analysis is made using either two sample t-test or Wilcoxon's rank sum test.

SECONDARY OUTCOMES:
The variance in edema index between groups at weeks 4 and 8, compared to the baseline | Edema indexs (ECW/TBW) are measured at week 4, 8, 12 of treatment.
  Descriptive statistics (number of observation subjects, mean, standard deviation, median, minimum, maximum) are summarized by treatment group. Depending on whether there is a difference in the variance between treatment groups (S-amlodipine group, Amlodipine group) that satisfies the normality assumption, analysis is made using either two sample t-test or Wilcoxon's rank sum test.
The variance in ankle size (mean size of both ankles using a medical tape measure) between groups at weeks 4, 8, and 12, compared to the baseline. | Ankel sizes are measured in at week 4, 8, and 12 of treatment.
  Mean size of both anckles are tape-measured using medical tape.
The variance in edema index (extracellular moisture per site/water per site) by site (body, right arm, left arm, trunk, right leg, left leg) between groups at weeks 4, 8, and 12, compared to the baseline. | Edema indexs (ECW/TBW) by site (body, right arm, left arm, trunk, right leg, left leg) are measured at the week 4, 8, and 12 of treatment.
  Descriptive statistics (number of observation subjects, mean, standard deviation, median, minimum, maximum) are summarized by site(body, right arm, left arm, trunk, right leg, left leg) and treatment group. Depending on whether there is a difference in the variance between treatment groups (S-amlodipine group, Amlodipine group) that satisfies the normality assumption, analysis is made using either two sample t-test or Wilcoxon's rank sum test.
The variance in blood pressure between groups at weeks 4, 8, and 12, compared to the baseline. | Blood pressure are measured at week 4, 8, and 12 of treatment.
  Blood pressure is measured at five-minute intervals after a five-minute rest while seated; three measurements are made for one arm and the SBP and DBP values at each measurement are collected and calculated to derive the mean value.

CONTACTS AND LOCATIONS:
Overall Officials: Eung Ju Kim, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pathak L, Hiremath, Kerkar PG, Manade VG. Multicentric, clinical trial of S-Amlodipine 2.5 mg versus Amlodipine 5 mg in the treatment of mild to moderate hypertension--a randomized, double-blind clinical trial. J Assoc Physicians India. 2004 Mar;52:197-202. PMID 15636308
- [Background] Pedrinelli R, Dell'Omo G, Melillo E, Mariani M. Amlodipine, enalapril, and dependent leg edema in essential hypertension. Hypertension. 2000 Feb;35(2):621-5. doi: 10.1161/01.hyp.35.2.621. PMID 10679507
- [Background] Messerli FH. Vasodilatory edema: a common side effect of antihypertensive therapy. Curr Cardiol Rep. 2002 Nov;4(6):479-82. doi: 10.1007/s11886-002-0110-9. PMID 12379167
- [Background] Sener D, Halil M, Yavuz BB, Cankurtaran M, Ariogul S. Anasarca edema with amlodipine treatment. Ann Pharmacother. 2005 Apr;39(4):761-3. doi: 10.1345/aph.1E410. Epub 2005 Feb 22. PMID 15728328
- [Background] Brown NJ, Vaughan DE. Angiotensin-converting enzyme inhibitors. Circulation. 1998 Apr 14;97(14):1411-20. doi: 10.1161/01.cir.97.14.1411. PMID 9577953
- [Background] Elliott WJ, Meyer PM. Incident diabetes in clinical trials of antihypertensive drugs: a network meta-analysis. Lancet. 2007 Jan 20;369(9557):201-7. doi: 10.1016/S0140-6736(07)60108-1. PMID 17240286
- [Background] Makani H, Bangalore S, Romero J, Htyte N, Berrios RS, Makwana H, Messerli FH. Peripheral edema associated with calcium channel blockers: incidence and withdrawal rate--a meta-analysis of randomized trials. J Hypertens. 2011 Jul;29(7):1270-80. doi: 10.1097/HJH.0b013e3283472643. PMID 21558959
- [Background] Galappatthy P, Waniganayake YC, Sabeer MI, Wijethunga TJ, Galappatthy GK, Ekanayaka RA. Leg edema with (S)-amlodipine vs conventional amlodipine given in triple therapy for hypertension: a randomized double blind controlled clinical trial. BMC Cardiovasc Disord. 2016 Sep 1;16(1):168. doi: 10.1186/s12872-016-0350-z. PMID 27586538
- [Background] Liu F, Qiu M, Zhai SD. Tolerability and effectiveness of (S)-amlodipine compared with racemic amlodipine in hypertension: a systematic review and meta-analysis. Curr Ther Res Clin Exp. 2010 Feb;71(1):1-29. doi: 10.1016/j.curtheres.2010.02.005. PMID 24683248
- [Background] Kim SA, Park S, Chung N, Lim DS, Yang JY, Oh BH, Tahk SJ, Ahn TH. Efficacy and safety profiles of a new S(-)-amlodipine nicotinate formulation versus racemic amlodipine besylate in adult Korean patients with mild to moderate hypertension: an 8-week, multicenter, randomized, double-blind, double-dummy, parallel-group, phase III, noninferiority clinical trial. Clin Ther. 2008 May;30(5):845-57. doi: 10.1016/j.clinthera.2008.05.013. PMID 18555932
- [Background] Schoeller DA, Alon A, Manekas D, Mixson LA, Lasseter KC, Noonan GP, Bolognese JA, Heymsfield SB, Beals CR, Nunes I. Segmental bioimpedance for measuring amlodipine-induced pedal edema: a placebo-controlled study. Clin Ther. 2012 Mar;34(3):580-92. doi: 10.1016/j.clinthera.2012.01.018. Epub 2012 Mar 3. PMID 22385927